CLINICAL TRIAL: NCT00701428
Title: Phase 4 Study of Losartan in Hypertensive Men and Women With Obstructive Sleep Apnea Before and After Continuous Positive Airway Pressure (CPAP) Treatment
Brief Title: Losartan in Hypertensive Men and Women With Sleep Apnea Before and on Continuous Positive Airway Pressure (CPAP) Treatment
Acronym: LosartanPAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Skaraborg Hospital (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Yuksel Peker, MD, PhD, Associate Professor, Skaraborg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGSKAS-12916; FoU Sweden, nr 8751
Record Dates: First submitted 2008-06-13; First posted 2008-06-19 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Hypertension; Sleep Apnea
Keywords: Hypertension; Sleep Apnea; Angiotensin II antagonist; CPAP
MeSH Terms: conditions — Hypertension; Sleep Apnea Syndromes | interventions — Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Hypertensive Men and Women Without OSA on Losartan (n=30)
  Interventions: Drug: Losartan
- 2 (Active Comparator): Hypertensive Men and Women With OSA on Losartan (n=30)
  Interventions: Drug: Losartan
- 3 (Experimental): Hypertensive Men and Women with OSA on Losartan and CPAP (n=30)
  Interventions: Drug: Losartan; Other: CPAP

INTERVENTIONS:
Drug: Losartan — Losartan 50 mg daily during 6 + 6 weeks
  Other Names: Cozaar
Other: CPAP — CPAP during the second 6 week-period
  Other Names: Auto-CPAP
  Arms: 3

SUMMARY:
Obstructive sleep apnea (OSA) is a highly prevalent condition in hypertensive patients. The renin-angiotension-aldosterone-system (RAAS) has a central role in blood pressure control. An angiotensin-II-antagonist, Losartan, is an effective antihypertensive drug. However, some patients respond to this drug worse than the others, and it is a clinical praxis to either increase the dosage and/or add another drug. There is limited data regarding the impact of antihypertensive drugs in OSA patients, i.e., whether or not OSA may constitute the subgroup of therapy-resistent hypertensive patients. In the literature, there is no data, either, whether or not CPAP treatment may have an additive blood pressure lowering impact in this certain subgroup.

DETAILED DESCRIPTION:
OSA is a highly prevalent condition in hypertensive patients and the prevalence is even higher in patients with drug-resistant hypertension. The renin-angiotension-aldosterone-system (RAAS) has a central role in blood pressure control. An angiotensin-II-antagonist, Losartan, has an effective antihypertensive drug. However, some patients respond to this drug worse than the others, and it is a clinical praxis to either increase the dosage and/or add another drug. There is limited data regarding the impact of antihypertensive drugs in OSA patients, i.e., whether or not OSA may constitute the subgroup of therapy-resistent hypertensive patients. In the literature, there is no data, either, whether or not CPAP treatment may have an additive blood pressure lowering impact in this certain subgroup. The investigators will include 90 otherwise healthy, untreated hypertensive men and women(age 50-69 yrs, Body-Mass-Index <35 kg/m2; 60 patients with OSA, 30 non-OSA) as described above. Before start of treatment, fasting blood samples will be drawn regarding the neuroendocrine hormones (adrenaline, noradrenaline, plasma renin activity, angiotensin II,aldosterone, pro-BNP) and cardiovascular biomarkers (CRP,interleukines, cytokines). All subjects will start with Losartan 50 mg and 24 h- blood-pressure response and blood sample analysis will be compared between OSA and non-OSA subjects after 6 weeks of treatment. In the second 6-week period, all subjects will continue with Losartan while the half of the OSA group (n=30) will be randomized to CPAP and the other 30 patients will continue with Losartan only.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index <35 kg/m2
* Systolic Blood Pressure >=140 mmHg and/or Diastolic Blood Pressure >=95 mmHg
* No known clinical disease except hypertension
* No cardiovascular medication
* Apnea-Hypopnea Index < 5/h (no OSA), or Apnea Hypopnea Index >=15/h (OSA)

Exclusion Criteria:

* Manifest diabetes, liver- or kidney disease Signs of atrial fibrillation or former myocardial infarction at electrocardiogram

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-06; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
24 h blood pressure (mean blood pressure; mmHg) | Changes from Baseline in 24 h BP at 6 and 12 weeks, respectively

SECONDARY OUTCOMES:
Markers of sympathetic activity, RAAS-activity, cardiovascular biomarkers | Changes from Baseline in Biomarkers at 6 and 12 weeks, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Yuksel Peker, Prof., Principal Investigator — Göteborg University; Erik Thunström, PhD, Principal Investigator — Göteborg University
Locations (1):
- University of Gothenburg, Sahlgrenska Academy, Gothenburg, West Gotaland, Sweden

REFERENCES:
- [Result] Thunstrom E, Manhem K, Rosengren A, Peker Y. Blood Pressure Response to Losartan and Continuous Positive Airway Pressure in Hypertension and Obstructive Sleep Apnea. Am J Respir Crit Care Med. 2016 Feb 1;193(3):310-20. doi: 10.1164/rccm.201505-0998OC. PMID 26414380
- [Result] Thunstrom E, Manhem K, Yucel-Lindberg T, Rosengren A, Lindberg C, Peker Y. Neuroendocrine and Inflammatory Responses to Losartan and Continuous Positive Airway Pressure in Patients with Hypertension and Obstructive Sleep Apnea. A Randomized Controlled Trial. Ann Am Thorac Soc. 2016 Nov;13(11):2002-2011. doi: 10.1513/AnnalsATS.201602-126OC. PMID 27548072